CLINICAL TRIAL: NCT04422548
Title: Does AI-assisted Colonoscopy Improve Adenoma Detection in Screening Colonoscopy? A Multi-center Randomized Controlled
Brief Title: Does AI-assisted Colonoscopy Improve Adenoma Detection in Screening Colonoscopy?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joseph JY SUNG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AI-CLN Study_Protocol
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Screening Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assisted Group (Active Comparator)
  Interventions: Procedure: AI-assisted Colonoscopy
- Standard (Active Comparator)
  Interventions: Procedure: Standard Colonoscopy

INTERVENTIONS:
Procedure: AI-assisted Colonoscopy — This is a multi-center prospective randomized controlled study comparing real-time AI-assisted colonoscopy versus standard colonoscopy in a real-life setting.
  Arms: AI-assisted Group
Procedure: Standard Colonoscopy — Standard Colonoscopy
  Arms: Standard

SUMMARY:
To date, there is a lack of large-scale randomized controlled study using AI assistance in the detection of polyps/adenoma in a screening population. The correlation of fecal occult blood test (FIT or FOBT) and the advantage of AI-assisted colonoscopy has not been investigated. There is also a lack of information of the benefit of AI-assisted colonoscopy in experienced colonoscopist versus trainee/resident.

DETAILED DESCRIPTION:
There are several studies showing that AI-assisted colonoscopy can help in identifying and characterizing polyps found on colonoscopy.

* Byrne et al demonstrated that their AI model for real-time assessment of endoscopic video images of colorectal polyp can differentiate between hyperplastic diminutive polyps vs adenomatous polyps with sensitivity of 98% and specificity of 83% (Byrne et al. GUT 2019)
* Urban et al designed and trained deep CNNs to detect polyps in archived video with a ROC curve of 0.991 and accuracy of 96.4%. The total number of polyps identified is significantly higher but mainly in the small (1-3mm and 4-6mm polyps) (Urban et al. Gastroenterol 2018)
* Wang et al conducted an open, non-blinded trial consecutive patients (n=1058) prospectively randomized to undergo diagnostic colonoscopy with or without AI assistance. They found that AI system increased ADR from 20.3% to 29.1% and the mean number of adenomas per patients from 0.31 to 0.53. This was due to a higher number of diminutive polyps found while there was no statistic difference in larger adenoma. (Wang et al. GUT 2019). In this study, they excluded patients with IBD, CRC and colorectal surgery. The patients presented with symptoms to hospital for investigation.

To date, there is a lack of large-scale randomized controlled study using AI assistance in the detection of polyps/adenoma in a screening population. The correlation of fecal occult blood test (FIT or FOBT) and the advantage of AI-assisted colonoscopy has not been investigated. There is also a lack of information of the benefit of AI-assisted colonoscopy in experienced colonoscopist versus trainee/resident.

ELIGIBILITY:
Inclusion Criteria

* Patients receiving colonoscopy screening
* Patients aged 45-75 years
* Both patients who have or have not done a FIT test and both FIT +ve and FIT -ve subjects

Exclusion Criteria

* Patients who have symptom(s) suggestive of colorectal diseases
* Patients who have a history of inflammatory bowel disease, colorectal cancer or polyposis syndrome (anaemia, bloody stool, tenesmus and obstructive symptoms)
* Patients who had colonoscopy or other investigation of colon and rectum in the past 10 years
* Patients who had surgery for colorectal diseases
* Patients who cannot tolerate bowel preparation or have suboptimal bowel preparations (Boston Bowel Preparation Scale)
* Cannot reach caecum
* Patients who are incompetent in giving informed consent

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2994 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-11-27 (Estimated); Study Completion 2020-11-27 (Estimated)

PRIMARY OUTCOMES:
Per-patient ADR in each group | 12 months
  For the AI-Assisted group, it is defined as the number of patients with at least 1 adenoma identified in the colon divided by the total number of patients in the AI-Assisted group.
Per-patient ADR in each group | 12 months
  For the Standard group, it is defined as the number of patients with at least 1 adenoma identified in the colon divided by the total number of patients in the Standard group.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu H, Tang RSY, Lam TYT, Zhao G, Lau JYW, Liu Y, Wu Q, Rong L, Xu W, Li X, Wong SH, Cai S, Wang J, Liu G, Ma T, Liang X, Mak JWY, Xu H, Yuan P, Cao T, Li F, Ye Z, Shutian Z, Sung JJY. Artificial Intelligence-Assisted Colonoscopy for Colorectal Cancer Screening: A Multicenter Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2023 Feb;21(2):337-346.e3. doi: 10.1016/j.cgh.2022.07.006. Epub 2022 Jul 19. PMID 35863686